CLINICAL TRIAL: NCT05529173
Title: A Prospective Single-blind Placebo-controlled Trial to Establish the Efficacy and Tolerability of 10% Povidone-Iodine for Nasal S. Aureus and Methicillin Resistant S. Aureus (MRSA) Decolonization Among Patients Undergoing Same-day Surgery
Brief Title: Povidone-Iodine for Nasal Decolonization
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Dennis Grech, MD, Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro2021000468
Record Dates: First submitted 2022-09-01; First posted 2022-09-06 (Actual); Results first posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-10

CONDITIONS: Surgical Wound Infection; Preoperative Care; Methicillin-Resistant Staphylococcus Aureus
MeSH Terms: conditions — Surgical Wound Infection | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Patients are assigned to treatment group or placebo
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- treatment (Experimental): Application of Povidone-Iodine 10% prior to surgery to Nares
  Interventions: Drug: Povidone-Iodine 10%
- placebo (Placebo Comparator): Application of 0.9% Sodium Chloride (NaCl) solution prior to surgery to Nares
  Interventions: Drug: 0.9% NaCl Solution

INTERVENTIONS:
Drug: Povidone-Iodine 10% — Nasal swab stick application of Povidone-Iodine 10% prior to surgery
  Other Names: Profend
  Arms: treatment
Drug: 0.9% NaCl Solution — Nasal swab stick application of 0.9% NaCl Solution prior to surgery
  Other Names: Normal Saline (NS)
  Arms: placebo

SUMMARY:
To evaluate the efficacy and tolerability of 10% povidone-iodine in eliminating nasal carriage of Staphylococcus aureus and MRSA. To determine whether a more convenient, single-dose, pre-operative 10% povidone-iodine (PI) application is effective in reducing nasal carriage of S. aureus and MRSA. We expect a statistically significant decrease in S. aureus/MRSA colonization in nasal cultures taken perioperatively after intervention in patients who received pretreatment with PI as compared to patients who received normal saline (NS).

DETAILED DESCRIPTION:
This will be a prospective single-blinded randomized placebo-controlled trial of two applications of a nasal 10% Povidone Iodine (PI) solution used on the intranasal mucosal surfaces of each nostril in the preoperative holding area within 2 h prior to surgical incision compared with NS using the same technique. Both the PI and NS will be applied by rotating the swab over the intranasal mucosal surface for 15 seconds; this process will be performed twice for both nostrils, using a new swab for each application. Nasal cultures will be obtained prior to PI or NS application as well as intraoperatively 1 hour and 2 hours after first surgical incision. The primary study end point is the decrease in S. aureus/MRSA colony forming units (CFU) in nasal cultures taken within 2 hours after intervention in patients who presented with a positive preintervention nasal culture. A secondary endpoint is the presence or absence of surgical site infections within 30 days postoperatively

ELIGIBILITY:
Inclusion Criteria:

* community-based patients ages 18-80
* American Society of Anesthesiology (ASA) 1-3
* undergoing an outpatient surgery for at least 1 hour and up to 6 hours duration

Exclusion Criteria:

* pregnancy
* allergy to povidone-iodine
* infectious indication for surgery or preexisting known infection/wound
* immunocompromised state
* use of chemotherapy or steroids within 30 days prior to surgery
* use of antimicrobial therapy within 30 days prior to surgery
* surgeries where field avoidance prevents intraoperative access to the nares

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2023-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex Bekker, MD/PhD, Study Chair — Rutgers University
Locations (1):
- University Hospital, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kirby JP, Mazuski JE. Prevention of surgical site infection. Surg Clin North Am. 2009 Apr;89(2):365-89, viii. doi: 10.1016/j.suc.2009.01.001. PMID 19281889
- [Background] Davis GB, Peric M, Chan LS, Wong AK, Sener SF. Identifying risk factors for surgical site infections in mastectomy patients using the National Surgical Quality Improvement Program database. Am J Surg. 2013 Feb;205(2):194-9. doi: 10.1016/j.amjsurg.2012.05.007. Epub 2012 Aug 31. PMID 22944390
- [Background] Craft RO, Damjanovic B, Colwell AS. Evidence-based protocol for infection control in immediate implant-based breast reconstruction. Ann Plast Surg. 2012 Oct;69(4):446-50. doi: 10.1097/SAP.0b013e31824a215a. PMID 22964685
- [Background] Kalra L, Camacho F, Whitener CJ, Du P, Miller M, Zalonis C, Julian KG. Risk of methicillin-resistant Staphylococcus aureus surgical site infection in patients with nasal MRSA colonization. Am J Infect Control. 2013 Dec;41(12):1253-7. doi: 10.1016/j.ajic.2013.05.021. Epub 2013 Aug 21. PMID 23973424
- [Background] Salih L, Tevell S, Mansson E, Nilsdotter-Augustinsson A, Hellmark B, Soderquist B. Staphylococcus epidermidis isolates from nares and prosthetic joint infections are mupirocin susceptible. J Bone Jt Infect. 2018 Jan 1;3(1):1-4. doi: 10.7150/jbji.22459. eCollection 2018. PMID 29291157

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment | Placebo
Started | 95 | 97
Completed | 88 | 91
Not Completed | 7 | 6
Not completed — Physician Decision | 3 | 6
Not completed — Sample shipment delay more than one day | 4 | 0

BASELINE CHARACTERISTICS:
Population: Nasal samples were analyzed for 88 participants randomized to the treatment group and 91 participants randomized to the placebo group.
Units Other Than Participants: Nasal samples
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Placebo | Total
Number analyzed (Participants) | 95 | 97 | 192
Number analyzed (Nasal samples) | 88 | 91 | 179
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 88 | 86 | 174
  >=65 years | 7 | 11 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.86 (14.97) | 47.27 (14.84) | 46.08 (14.92)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 49 | 51 | 100
  Male | 44 | 45 | 89
  Prefer not to identify | 0 | 1 | 1
  Unknown | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 38 | 46 | 84
  White Non-Hispanic | 12 | 13 | 25
  Asian | 2 | 4 | 6
  Hispanic or Latino | 37 | 31 | 68
  Other | 4 | 2 | 6
  Unknown | 2 | 1 | 3
Number of S. aureus/ MRSA colony-forming unit (CFU) per Sample [Median (Inter-Quartile Range); unit: CFU per sample] — Population: Row population differs from the overall as nasal samples of 7 participants from the treatment group and 6 from the placebo group were not analyzed due to shipment delay or other reasons.
  CFU per sample
    number analyzed (Participants) | 88 | 91 | 179
    Number of S. aureus CFU per Sample | 2500 [25 to 20350] | 2500 [526.5 to 31800] | 2500 [250 to 24775]
    Number of MRSA CFU per Sample | 125.5 [25 to 2500] | 25 [25 to 2500] | 51.8 [25 to 2500]

OUTCOME MEASURES:

1. Primary Outcome: Change in S. Aureus/MRSA Colony Forming Units (CFU) in Nasal Swab Specimen After Treatment in Patients Who Presented With a Positive for S. Aureus/MRSA Pre-interventional Nasal Swab Specimen.
Description: The difference in a number of S. aureus/MRSA CFU in nasal swab specimens between before and after the study drug/placebo application in patients with a positive for S. aureus/MRSA pre-interventional nasal swab specimen. The change (Δ) is calculated as the value at the baseline time point minus the value at the later time point. Positive values represent a decrease in CFU, whereas negative values represent an increase in CFU.
Time Frame: 1, 2, and 3 hours after application of Povidone-Iodine or saline solution
Population: Nasal samples (NS) taken from 42 participants out of 95 assigned to the treatment group, and 47 out of 97 assigned to the placebo group that tested positive for S. aureus before the intervention were analyzed at every following time point: 1, 2, and 3 hours after the intervention (AI).
  NS taken from 32 participants out of 95 assigned to the treatment group, and 35 out of 97 assigned to the placebo group were positive for MRSA at baseline and were analyzed for MRSA at 1,2, and 3 hours AI.
Measure: Median (Inter-Quartile Range); unit: CFU per sample (∆)
Units Other Than Participants: nasal samples
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 42 | 47
Number analyzed (nasal samples) | 42 | 47
CFU per sample (∆)
  The difference in a number of S. aureus CFU between before and 1 hour after drug application | 12062.5 [2007.5 to 46023.6] | 737 [-29445 to 27850]
  The difference in a number of S. aureus CFU between before and 2 hours after drug applicatia | 12525 [815 to 61425] | 711.2 [-24411 to 58400]
  The difference in a number of S. aureus CFU between before and 3 hours after drug application | 12497 [1045.5 to 38075.1] | 4160 [-2481.5 to 82383]
  The difference in a number of MRSA CFU between before and 1 hour after drug application: number analyzed (Participants) | 32 | 35
  The difference in a number of MRSA CFU between before and 1 hour after drug application: number analyzed (nasal samples) | 32 | 35
  The difference in a number of MRSA CFU between before and 1 hour after drug application | 2904.8 [349.3 to 18175] | 360 [-2434.1 to 3126.7]
  The difference in a number of MRSA CFU between before and 2 hours after drug application: number analyzed (Participants) | 32 | 35
  The difference in a number of MRSA CFU between before and 2 hours after drug application: number analyzed (nasal samples) | 32 | 35
  The difference in a number of MRSA CFU between before and 2 hours after drug application | 2457 [254.5 to 18175] | 412 [-7024.1 to 4811]
  The difference in a number of MRSA CFU between before and 3 hours after drug application: number analyzed (Participants) | 32 | 35
  The difference in a number of MRSA CFU between before and 3 hours after drug application: number analyzed (nasal samples) | 32 | 35
  The difference in a number of MRSA CFU between before and 3 hours after drug application | 2904.8 [349.3 to 18175] | 360 [-2434.1 to 3126.7]
Statistical Analysis 1: Comparison: Treatment vs Placebo; Test type: Other; p < 0.05, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Surgical Site Infections
Description: The presence of surgical site infections
Time Frame: at 7 and 30-day postoperative intervals
Population: Row population differs from the overall as the secondary outcome was analyzed for 88 out of 95 participants assigned to the treatment group and 91 out of 97 to the placebo group.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 88 | 91
Participants
  Confirmed surgical site infection in the first 7 days postoperatively | 0 | 1
  Confirmed surgical site infection up to 30±4 days postoperatively | 1 | 6

ADVERSE EVENTS:
Time Frame: From the time the patient signs the Informed Consent Form for 24 hours or until discharge from the hospital, whatever comes first, an average of 12 hours
Arm/Group | Treatment | Placebo
All-Cause Mortality (participants affected / at risk) | 0/95 | 0/97
Serious Adverse Events (participants affected / at risk) | 0/95 | 0/97
Other Adverse Events (participants affected / at risk) | 2/95 | 0/97
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=95) | Placebo (N=97)
nasal irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — itching
nasal irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — running nose

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-06): https://cdn.clinicaltrials.gov/large-docs/73/NCT05529173/Prot_SAP_002.pdf
  • Informed Consent Form (2023-06-28): https://cdn.clinicaltrials.gov/large-docs/73/NCT05529173/ICF_000.pdf